CLINICAL TRIAL: NCT03676036
Title: A Prospective, Randomised, Vehicle-Controlled, Double-Blind, Exploratory Clinical Trial To Assess The Efficacy And Steroid Sparing Potential Of DGLA Cream Topically Applied To Patients With Moderate To Severe Atopic Dermatitis
Brief Title: Efficacy and Steroid Sparing Potential Study of DGLA Cream in Patients With Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DS Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DS107E-04
Record Dates: First submitted 2018-01-30; First posted 2018-09-18 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- DS107E and Steroid (Experimental): First 7 days: Steroid taken topically once a day and DS107E taken once a day Next 28 days: DS107E taken topically twice a day
  Interventions: Drug: DS107E
- Vehicle and Steroid (Placebo Comparator): First 7 days: Steroid taken topically once a day and Vehicle taken once a day Next 28 days: Vehicle taken topically twice a day
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: DS107E
  Other Names: Mometasone Furoate
  Arms: DS107E and Steroid
Drug: Vehicle
  Other Names: Mometasone Furoate
  Arms: Vehicle and Steroid

SUMMARY:
This study will investigate the steroid sparing potential of DS107E to vehicle in patients with moderate to severe atopic dermatitis.

DS107E or vehicle will be topically administered with a steroid twice a day for the first 7 days. For the following 28 days DS107E or vehicle will be topically administered twice a day.

This study will enrol approximately 40 adult patients.

DETAILED DESCRIPTION:
Subjects will come to the clinic on 7 occasions: Screening, Baseline, Day 7, Day 14, Day 21, Day 35 (End of Treatment) and Day 42 (Follow-up). The primary efficacy variable will be EASI (Eczema Area and Severity Index). The secondary efficacy variables will be EASI, IGA (Investigators Global Assessment), SCORAD (SCORing Atopic Dermatitis), Target Lesion Score, VAS (Visual Analogue Scale), Skin Tolerability, DLQI (Dermatology Life Quality Index), Erythema, TEWL (Transepidermal Water Loss) and Time to Rescue Medication.

ELIGIBILITY:
Inclusion Criteria:

* Female and male volunteers aged 18-65 who are willing to give written informed consent.
* Diagnosis of atopic dermatitis (> 6 months) according to the Hanifin and Raika Criteria;
* Presence of at least 2 moderate to severe (target lesion score</=8) inflammatory lesions of comparable severity, erythema >/= 2
* Patients with moderate to severe atopic dermatitis (IGA=3-4)
* A body surface area score of less than 20%

Exclusion Criteria:

* Clinically significant impairment of renal or hepatic function.
* Other skin conditions that might interfere with atopic dermatitis diagnosis and/or evaluation (such as psoriasis or current viral, bacterial and fungal skin infections).
* History of intolerance to any ingredient in DS107E DGLA cream or Vehicle or intolerance to any ingredient in Ecural®(Mometasone furoate 0.1%). Of note, any intolerance to PHB ester (benzoate, parabens) or soy or it's cross-allergen peanut, as these are ingredients of DS107E.
* Use of biologics 3 months prior to start of treatment/ Day 0 visit (baseline), or 5 half-lives (whichever is longer).
* Use of systemic treatments (other than biologics) that could affect atopic dermatitis less than 4 weeks prior to baseline visit (Day 0), e.g. retinoids, calcineurin inhibitors, methotrexate, cyclosporine, hydroxycarbamide (hydroxyurea), azathioprine and oral/injectable corticosteroids; Intranasal corticosteroids and inhaled corticosteroids for stable medical conditions are allowed.
* Treatment with any experimental drug within 30 days prior to Day 0 visit (baseline), or 5 half lives (whichever is longer).
* Excessive sun exposure, use of tanning booths or other ultraviolet (UV) light sources 4 weeks prior to Day 0 visit (baseline) and/or is planning a trip to sunny climate or to use tanning booths or other UV sources between screening and follow-up visits.
* Use of any topical medicated treatment for atopic dermatitis 2 weeks prior to start of treatment/Day 0 visit (baseline), including but not limited to, topical corticosteroids, calcineurin inhibitors, tars, bleach, antimicrobials and bleach baths.
* Use of topical products containing ceramides 2 weeks prior to Day 0. Topical products that do not contain ceramides are allowed.
* Use of anti-histamines for atopic dermatitis within 2 weeks of baseline.
* Medical history of chronic infectious disease (e.g., hepatitis B, hepatitis C or infection with human immunodeficiency virus).
* History of clinically significant drug or alcohol abuse in the last year prior to Day 0 (baseline).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Eczema Area and Severity Index (EASI) | 5 weeks
  Four anatomic sites - head/neck, upper extremities, trunk and lower extremities - are assessed for erythema, induration (papules), excoriation and lichenification as seen on the day of the examination. The severity of each sign is assessed using a 4-point scale

SECONDARY OUTCOMES:
Eczema Area and Severity Index (EASI) | Days 7, 14, 21 and 35
  Four anatomic sites - head/neck, upper extremities, trunk and lower extremities - are assessed for erythema, induration (papules), excoriation and lichenification as seen on the day of the examination. The severity of each sign is assessed using a 4-point scale
Investigator Global Assessment (IGA) | Days 7, 14, 21 and 35
  The IGA scale awards a score of 0-4 from clear to severe disease. IGA uses clinical characteristics of erythema, infiltration, population and oozing as scoring guidelines for the overall severity assessment.
SCORing Atopic Dermatitis | Days 7, 14, 21 and 35
  Six items (erythema, edema/papulation, oozing/crusts, excoriation, lichenification, and dryness) are selected to evaluate the AD severity. The intensity of each item is graded using a 4-point scale.
Target Lesion Score | Days 7, 14, 21 and 35
  Moderate to severe target lesions will be graded for erythema, induration, excoriation and lichenification using local SCORAD scales.
Visual Analogue Scale (VAS) | Days 7, 14, 21 and 35
  11 points scale to assess pruritus
Skin Tolerability | Days 7, 14, 21 and 35
  Skin tolerability will be self-assessed by the subjects using a questionnaire.
Dermatology Life Quality Index | Days 7, 14, 21 and 35
  The DLQI is a simple 10-question validated questionnaire which will be completed at each visit.
Erythema | Days 7, 14, 21 and 35
  Erythema will be assessed with the skin Colorimeter CL 400
Transepidermal Water Loss | Days 7, 14, 21 and 35
  Measures the effect on skin barrier function.
Time to Rescue Medication | 5 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- DS Biopharma Investigational Site, Lübeck, Germany